CLINICAL TRIAL: NCT03595969
Title: Association Between Mitochondrial DNA Content and Risk of Acute Leukemia in Young Adult
Brief Title: Association Between Mitochondrial DNA Content and Risk of Acute Leukemia
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Lipeng Liu, M.D., Chinese Academy of Medical Sciences
Other Study IDs: YL2018070101
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Lymphoblastic Leukemia in Children
Keywords: mitochondrial DNA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- acute leukemia group: 150 patients were recruited, who have diagnosed with acute leukemia by bone marrow biopsy
  Interventions: Diagnostic Test: Relative copy number of mitochondrial DNA
- Control group: The 50 healthy controls without previous cancer history were recruited from individuals who visited investigator's hospital for physical examination during the same time period as the case enrollment.
  Interventions: Diagnostic Test: Relative copy number of mitochondrial DNA

INTERVENTIONS:
Diagnostic Test: Relative copy number of mitochondrial DNA — Mitochondria are responsible for multiple cellular functions including regulation of energy production, modulation of oxidation-reduction status, generation of reactive oxygen species and apoptosis. Each mitochondrion possesses multiple copies of a mitochondrial genome comprised of independently replicating double stranded DNA (mtDNA).

SUMMARY:
Compelling epidemiological evidence indicates that alterations of mitochondrial DNA, including mutations and abnormal content of mitochondrial DNA (mtDNA), are associated with the initiation and development of acute lymphoblastic leukemia (ALL).The aim of this study was to explore association between mtDNA content in peripheral blood cells could be used as a risk predictor for ALL.

ELIGIBILITY:
Inclusion Criteria:

* 1.histological confirmed chronic lymphocytic leukemia; 2.preparing for chemotherapy; 3.no preoperative anticancer treatment.

Exclusion Criteria:

* 1.history of other malignancy; 2.blood transfusion within one month or prior bone marrow transplantation; 3.patients who reluctant to sign informed consent.

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of 150 eligible chronic lymphocytic leukemia patients were anticipated to include in this study. Moreover, 50 healthy controls without previous cancer history were also recruited from individuals who visited investigator's hospital for physical examination during the same time period.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Relative copy number of mitochondrial DNA | From date of admission until the date of discharging from hospital, assessed up to 5 days
  The ratio of mitochondrial DNA contents to hemoglobin contents was calculated for each sample from standard curves. After that, the ratio for each sample was normalized to a calibrator DNA in order to standardize between different runs, and then defined as the measurement of relative mtDNA contents.Relative expression of mtDNA were measured in young adults suffered from chronic lymphocytic leukemiawhen compared with control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiao-Fan Zhu, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No